CLINICAL TRIAL: NCT05794100
Title: Evaluating the Impact of Different Sugar Replacer Combinations on Gastrointestinal Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KBE062 / BIO-2110
Record Dates: First submitted 2021-11-25; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Tolerance; Healthy Population
Keywords: Sugar replacer; Gastrointestinal symptoms; GITQ; BHD-BSS; Acute; microbiota

STUDY DESIGN:
Intervention Model Description: Each subject will be allocated to a sequence of consumption of the 10 different products
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Products have been produced with different shapes and with very close texture, colors and taste. They are packaged in individual portion bags labeled "Product 1" to "Product 10".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Test 1 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + Allulose provided at a dose of 1 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 2 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + Allulose provided at a dose of 1.75 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 3 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + Allulose provided at a dose of 2.5 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 4 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + FOS provided at a dose of 1 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 5 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + FOS provided at a dose of 1.75 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 6 (Active Comparator): No-sugar chewable candy containing Soluble Corn Fiber + Inulin + FOS provided at a dose of 2.5 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 7 (Active Comparator): No-sugar chewable candy containing Maltitol + Polydextrose provided at a dose of 1 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 8 (Active Comparator): No-sugar chewable candy containing Maltitol + Polydextrose provided at a dose of 1.75 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 9 (Active Comparator): No-sugar chewable candy containing Maltitol + Polydextrose provided at a dose of 2.5 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator
- Test 10 (Placebo Comparator): Control chewable candy made with sugar and provided at a dose of 1 serving equivalent
  Interventions: Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator

INTERVENTIONS:
Other: Acute intake of one of the products (active comparator 1 to 9) or Placebo comparator — One pack of each product (1 to 10) will be consumed on a separate occasion
  Other Names: No sugar chewable candies

SUMMARY:
This study is a randomized, double-blind, crossover trial aiming at evaluating the gastrointestinal tolerance of 3 sugar replacers mixes at 3 different doses. The investigators will also try to understand the factors that could explain the presence or absence of symptoms

DETAILED DESCRIPTION:
This study is a randomized, double-blind, crossover trial with 23 visits consisting of one screening visit, one baseline visit, and 21 study visits (10 test periods each consisting of 2 test visits and one drop-off visit) across 11 weeks. For this study, 60 generally healthy subjects will be randomized to a test sequence and will consume one control product and nine test products over the course of the study. Before consumption of any study products, breath hydrogen lactulose assessment and collection of stool samples for microbiome analysis will be completed. Additionally, midway through the study, data will be reviewed in a blinded manner and a stool sample will be collected from a subset of 30 subjects for in vitro fermentation tests. Gastrointestinal symptoms and stool information will be collected using the Gastrointestinal Tolerance Questionnaire (GITQ) and Bowel Habit Diary with Bristol Stool Scale (BHD-BSS). The GITQ and BHD-BSS will be administered for 3 days and 7 days prior to study product consumption, respectively. Additionally, the GITQ and BHD-BSS will be collected throughout the day of study product consumption and the 2 days after product consumption. 24-h urine samples will be collected after study product consumption for urinary allulose analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-55 years of age, inclusive at Visit 1 (Day -11).
2. BMI of 18.5 to 32.0 kg/m2, inclusive, at Visit 1 (Day -11).
3. Have normal bowel movement habit (<3 bowel movements/d to >2 bowel movements/week) based on the BHD-BSS collected at Visit 2 (Day -4).
4. Consumes fiber at an amount no more than the average American diet [based on consumption of high-fiber containing plant-based foods (e.g., fruits, vegetables, legumes, pulses, nuts, and products labeled as good or excellent sources of fiber)].
5. Smokes 10 cigarettes or less in a day and has no plan to change nicotine habits during the study period.
6. Non-user or former users (cessation ≥12 mo) of any marijuana or hemp products and has no plans to use marijuana or hemp products during the study period.
7. Willing to maintain habitual dietary, lifestyle, and physical activity (with exceptions per study instructions) throughout the trial and willing to adhere to dietary, lifestyle, and physical activity requirements of the study.
8. Willing to limit alcohol consumption to ≤3 standard drinks/d and ≤7 standard drinks/week throughout the trial.
9. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
10. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Moderate or severe GI symptoms or 3-d total score of >2 for any individual GI symptom based on the baseline GITQ collected at Visit 2 (Day -4). Mild burping and/or flatulence totaling a 3-d score of >2 is acceptable.
2. Has a clinically significant GI-related reaction towards GI symptom-causing foods (e.g., beans and legumes, vegetables high in inulin, sodas or fruit drinks, sugar alcohols, inulin, fructooligosaccharides, gluten, and dairy products [see Appendix 3]) as judged by the Clinical Investigator.
3. Female subjects who typically experience change in GI symptoms or bowel habits (e.g., increased or decreased laxation, bloating, abdominal cramping) at the time of menstruation. Subjects with these issues may be included if they are able to reliably predict the onset and duration of their menstruation-related symptoms (e.g., always occur only during the first two days of menses), in the judgment of the Clinical Investigator. Test visits will be scheduled around menses.
4. Female subjects who is unwilling to wear a tampon during the collection of the 24-h urine samples when these collections occur during the time of menstruation.
5. Abnormal laboratory test results of clinical significance at Visit 1 (Day -11), at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to Visit 2 (Day -4), for subjects with abnormal laboratory test results.
6. Clinically important GI condition that would potentially interfere with the evaluation of the study products (e.g., inflammatory bowel disease, irritable bowel syndrome, gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies).
7. Recent (within 2 weeks of Visit 1; Day -11) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥3 loose or liquid stools/d).
8. Self-reported history (within 6 weeks of Visit 1; Day -11) of constipation or diarrhea at the discretion of the Clinical Investigator.
9. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
10. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -11). One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Day -11), in the judgment of the Clinical Investigator. If taken, the repeat blood pressure measurement will be used to determine eligibility. Stable use of hypertension medication is allowed [defined as no change in medication regimen within the 3 mo prior to Visit 1 (Day -11)].
11. Any known food allergy as well as intolerance or sensitivity to study product ingredients (Appendix 13).
12. Extreme dietary habits or physical activity patterns at the discretion of the Clinical Investigator.
13. History or presence of cancer in the prior 2 y, except for non-melanoma skin cancer.
14. Major trauma or any other surgical event within 3 mo of Visit 1 (Day -11).
15. Signs or symptoms of an active infection of clinical relevance within 5 d of Visit 1 (Day -11). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 d prior to Visit 1 (Day -11)*
16. Weight loss or gain > 4.5 kg in the 3 mo prior to Visit 1 (Day -11).
17. Currently or planning to be on a weight loss regimen during the study.
18. Antibiotic, antifungal, or antiparasitic use within 3 mo of Visit 1 (Day -11) and throughout the study period.
19. Use of steroids within 1 mo of Visit 1 (Day -11) and throughout the study period. Use of nasal and non-prescription topical treatments is allowed.
20. Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDS) within 1 mo of Visit 1 (Day -11).
21. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to prebiotics or probiotics, laxatives, enemas, fiber supplements and/or suppositories, antacids, anti-diarrheal agents, and/or anti-spasmodic within 3 weeks of Visit 1 (Day -11). Standard multivitamin and mineral supplements are allowed.
22. Participated in endoscopy or endoscopy preparation within 3 mo prior to Visit 1 (Day -11).
23. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Day -11).
24. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Subjects who are pregnant during the study will be discontinued.
25. Recent history (within 12 mo of screening; Visit 1; Day -11) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks/week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
26. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in area under the curve (AUC) of the composite Gastrointestinal symptom score of each test product versus control | AUC between 0 to 48 hours after intake of products
  AUC of the composite Gastrointestinal symptoms score based on GITQ (gastro-intestinal tolerance questionnaire)

SECONDARY OUTCOMES:
Difference in the continuous AUC of the composite GI symptom score between doses within each formulation | AUC between 0 to 48 hours after intake of products
  Area under the curve (AUC) of the composite GI symptoms score based on GITQ (gastro-intestinal tolerance questionnaire)
Difference in the continuous AUC of the composite GI symptom score between formulations within each dose | AUC between 0 to 48 hours after intake of products
  AUC of the composite GI symptoms score based on GITQ
Difference in the continuous AUC for each individual GI symptom score of test products as compared to control, dose within each formulation, and formulation within each dose | AUC between 0 to 48 hours after intake of products
  AUC of the composite GI symptoms score based on GITQ (gastro-intestinal tolerance questionnaire)
Proportion of subjects who have a composite GI symptom score larger than 1 at each measured time point | AUC between 0 to 48 hours after intake of products
  AUC of the composite GI symptoms score based on GITQ (gastro-intestinal tolerance questionnaire)
Proportion of subjects with diarrhea based on BHD-BSS (Bowel Habit Diary - Brictol Stool Scale) | Evaluation over 24 hours following intake of products
  diarrhea
Proportion of subjects that report any (score >0) or moderate-to-severe (score >1) symptom at each measured time point for each individual outcome | Evaluation performed at time 0, 120, 240, 360, 600 minutes and 24 and 48 hours
  Individual GI symptoms from GITQ (gastro-intestinal tolerance questionnaire)
Summary of the maximum detected score for each individual GI symptom | Evaluation performed at time 0, 120, 240, 360, 600 minutes and 24 and 48 hours
  Individual GI symptoms from GITQ (gastro-intestinal tolerance questionnaire)
Summary of the time of the maximum detected score for each individual symptom | Evaluation performed at time 0, 120, 240, 360, 600 minutes and 24 and 48 hours
  Individual GI symptoms from GITQ (gastro-intestinal tolerance questionnaire)
Proportion of subjects that report any (score >0) or moderate-to-severe (score >1) bothersome loose stools on the GITQ at each measured time point | Evaluation performed at time 0, 120, 240, 360, 600 minutes and 24 and 48 hours
  Loose stools from BHD-BSS (Bowel Habit Diary - Brictol Stool Scale)
Difference between test and control products, between dose within each formulation, and between formulation within each dose for all parameters of the BHD-BSS (Bowel Habit Diary - Brictol Stool Scale) | At each bowel movement over 48 hours
  Bowel movment characteristics from BHD-BSS (Bowel Habit Diary - Brictol Stool Scale)
Urinary allulose | Collect over 24 hours
  Difference between test and control products, between dose (number of servings) within each formulation, and between formulation within each dose on urinary Allulose
Gut Microbiota composition | Baseline
  Microbial composition by sequencing
Correlation analyses between microbiota composition and GITQ individual parameters | AUC 0 to 48 hours for composite scores and evaluations performed at time 0, 120, 240, 360, 600 minutes and 24 and 48 hours
  Mechanism of action

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Kelley, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No